CLINICAL TRIAL: NCT02937051
Title: Effects of Cigar Flavors on Measures of Abuse Liability Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20007848; R03DA043005 (NIH)
Record Dates: First submitted 2016-09-06; First posted 2016-10-18 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Tobacco Products
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Own Brand Cigarette Condition (Active Comparator)
  Interventions: Other: Tobacco product administration and assessment
- Original-flavor Black&Mild cigar (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- Apple-flavor Black&Mild cigar (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- Cream-flavor Black&Mild cigar (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- Wine-flavor Black&Mild cigar (Experimental)
  Interventions: Other: Tobacco product administration and assessment

INTERVENTIONS:
Other: Tobacco product administration and assessment — two bouts of 10 puffs of a tobacco product with a 30-second interpuff interval separated by 60 minutes; preceded and followed by physiological, subjective and topography assessment

SUMMARY:
This study involves 25 current young adult combustible tobacco cigarette (CTC) smokers who will complete 5 Latin square ordered, within-subject, laboratory conditions that differ by the tobacco product smoked:

1. own-brand CTC (positive control),
2. original-flavored Black & Mild (B&M) cigar,
3. apple-flavored B&M cigar,
4. cream-flavored B&M cigar, and
5. wine-flavored B&M cigar.

ELIGIBILITY:
Inclusion Criteria:

* To be included, participants must be healthy, as determined by self-report and heart rate/blood pressure (HR/BP) check, between the ages of 18-25, and willing to provide informed consent.
* They must agree to attend the lab and abstain from tobacco/nicotine as required, to use the designated products, and to follow the study protocol.
* Participants must also be regular CTC smokers (≥5 cigarettes/day for past 3 months) naïve to cigar products (smoked no more than 10 cigar products of any type in lifetime) who can provide a semi-quantitative urine cotinine result of ≥3 at screening (NicAlert test).

Exclusion Criteria:

* Individuals with a self-reported history of chronic diseases or psychiatric conditions will be excluded.
* Other exclusion criteria are: history of or active cardiovascular disease, current oral health problems or injuries, low/high BP, seizures, regular prescription medication use (other than vitamins or birth control), and past month use of cocaine, opioids, benzodiazepines, and methamphetamine (self-report).
* Individuals who report using marijuana or alcohol >20 days in the past 30 or interest in quitting CTC use within the next 30 days will also be excluded.
* Women will be excluded if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Change in saliva nicotine concentration | Saliva will be collected at baseline before the first product administration, at 10 min following each product administration, and 55 min following the first product administration (baseline for the second product administration).
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Change in breakpoint from two behavioral choice tasks (Cigarette Purchase Task, Multiple Choice Procedure) | A behavioral choice task (cigarette purchase cask) will be completed at baseline before the first product administration, 5, 15, 30, and 45 min following each bout. 45 min after the second bout, the multiple choice procedure will be administered.
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Change in Addiction Research Center Inventory subjective abuse liability | Subjective measures of abuse liability will be collected at baseline before the first product administration, 5, 15, 30, and 45 min following each bout.
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Change in Direct Effects of Nicotine and Tobacco Scale subjective abuse liability | Subjective measures of abuse liability will be collected at baseline before the first product administration, 5, 15, 30, and 45 min following each bout.
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Change in Tobacco Abstinence Symptoms and Drug Effects subjective abuse liability | Subjective measures of abuse liability will be collected at baseline before the first product administration, 5, 15, 30, and 45 min following each bout.
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).

SECONDARY OUTCOMES:
Expired air carbon monoxide | Expired air carbon monoxide measurement will occur at baseline before the first product administration, 15 minutes following each bout, 55 min following the first product administration (baseline for the second product administration).
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Heart rate | Heart rate will be recorded at one second intervals from session onset (minute zero of session) through minute 155 of the session (end of session).
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration.Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Blood pressure | Blood pressure will be recorded at 5 minute intervals from from session onset (minute zero of session) through minute 155 of the session (end of session).
  Each participant will attend 5 study sessions, each study session will include two bouts of product administration.Product administration will consist of 10 puffs with a 30-second interpuff interval (IPI; puff number and IPI will be directed and monitored by staff).
Puff Volume (ml) | Puff Volume will be measured in seconds for each puff during product administration (10 puffs with a 30-second interpuff interval directed and monitored by staff)
  The instrument senses flow-induced pressure drop across an orifice that is incorporated into the mouthpiece. Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Puff Volume and Puff Duration will be used to calculate measures of Puff Flow Rate (Puff Volume/Puff Duration) and Total Puff Volume (Puff Volume per puff x 10 puffs).
Puff Duration (seconds) | Puff Duration will be measured in seconds for each puff during product administration (10 puffs with a 30-second interpuff interval directed and monitored by staff)
  The instrument senses flow-induced pressure drop across an orifice that is incorporated into the mouthpiece. Each participant will attend 5 study sessions, each study session will include two bouts of product administration. Puff Volume and Puff Duration will be used to calculate measures of Puff Flow Rate (Puff Volume/Puff Duration) and Total Puff Volume (Puff Volume per puff x 10 puffs).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Barnes, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Behavioral Health Research Laboratory, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Once appropriate, a completely de-identified data set will be created that obfuscates any variable that might potentially be used to identify an individual study participant. In accordance with HIPAA definitions for public data sharing, the investigators will use standard acceptable processes that include removal of identifiers, translation of dates and ages to delta time values, assignment of random study identifiers, and any other methods acceptable at that time. A data sharing agreement will be required for release of any data. Individuals requesting a copy of study data will need to submit a detailed research plan that includes the purpose of the proposed research, the variables required, the duration of the analysis phase, IRB approval with FWA information, investigator training in human subjects, and other approvals specific to the individual datasets.

REFERENCES:
- [Derived] Wall CS, Bono RS, Lester RC, Hoetger C, Lipato T, Guy MC, Eissenberg TE, Bickel WK, Barnes AJ, Cobb CO. Triangulating abuse liability assessment for flavoured cigar products using physiological, behavioural economic and subjective assessments: a within-subjects clinical laboratory protocol. BMJ Open. 2018 Oct 10;8(10):e023850. doi: 10.1136/bmjopen-2018-023850. PMID 30309993

DOCUMENTS (1):
  • Informed Consent Form (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT02937051/ICF_001.pdf